CLINICAL TRIAL: NCT04371042
Title: PROtocol of Metabolic and Cryptogenic livEr Disease regisTry for intEgration of Omic Studies
Acronym: PROMETEO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 2576
Record Dates: First submitted 2020-01-23; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-01

CONDITIONS: NAFLD - Nonalcoholic Fatty Liver Disease; Diabetes; Obesity; Metabolic Syndrome; Cirrhosis; Liver Cancer; NASH - Nonalcoholic Steatohepatitis; HCC - Hepatocellular Carcinoma; Fatty Liver
Keywords: NAFLD; NASH; NON-ALCHOLIC; LIVER; CIRRHOSIS; HEPATOCELLULAR CARCINOMA
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus; Obesity; Metabolic Syndrome; Fibrosis; Liver Neoplasms; Carcinoma, Hepatocellular; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Clinical data will be collected in the electronic form at baseline and thereafter on an annual basis.
  In the prospective project, biological sample (DNA, RNA, sera or whole blood; urine, feces, bile and liver tissues) are collected, only on a voluntary basis, at the time of recruitment and follow-up and stored at the biobank facility XBIOGEM at Fondazione Policlinico Univ. A. Gemelli IRCCS in Rome
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aim of the study is to set up an observational cohort with NAFLD (Non-alcoholic fatty liver disease) at different stage of disease (from simple steatosis to cirrhosis and/or HCC-Hepatocellular carcinoma) and for comparative purpose a cohort of subjects with diabetes and/or obesity and/or other risk factors (i.e. psoriasis, IBD (inflammatory bowel disease), dyslipidemia) without NAFLD in order to have a clinical phenotypical characterization and the collection of biological specimens.

We will collect clinical data, biological samples and imaging results in order to perform future cross-sectional studies and/or longitudinal studies for elucidating pathways of the disease and develop and validate biomarkers for diagnosis, prognosis and monitoring liver disease and comorbidities in order to contribute to precision medicine in this field.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is characterized by the excessive accumulation of triglycerides in the liver and is often associated, in the absence of significant alcohol consumption, to insulin resistance and to the metabolic syndrome of which it shares the most frequent clinical manifestations (hypertension, dyslipidemia, visceral adiposity, glucose intolerance). Because of the pandemic spread of obesity and diabetes and by virtue of the best control of viral hepatitis, in western countries NAFLD is the most common cause of liver injury with prevalence that is around 20-30% of the general population.

NAFLD encompasses a broad spectrum of liver conditions associated with fat accumulation that ranges from benign fatty liver (FL), non-progressive liver fat accumulation to severe liver injury, cirrhosis, and liver failure. The histological signature ballooning degeneration (with or without Mallory bodies) and/or inflammation and/or fibrosis is typical of nonalcoholic steatohepatitis (NASH), that may progress to: i) cirrhosis and contribute to one category of cryptogenic cirrhosis (CC), in which steatosis may be present or absent; ii) hepatocellular carcinoma (HCC). Furthermore, the correct indication of subjects with significant fibrosis in the highest risk populations could also contribute to reducing the increasing prevalence of cirrhosis secondary to NAFLD as an indication to liver transplantation. Moreover, the expected impact of NAFLD and its complication on public health is quite impressive worldwide.

Hepatic steatosis is emerging as an early and common determinant of many of these diseases and co-morbidities, as reported also by our research group. Fatty liver, in fact, may cause lipid accumulation, inflammation, and oxidative stress at the hepatic level leading to NAFLD, and facilitating the occurrence of additional clinical co-morbidities by the activation of common molecular and cellular mechanisms. In fact, NAFLD is correlated to several metabolic diseases, such as Metabolic Syndrome (MetS), Cardiovascular Diseases (CVD), Chronic Kidney Disease (CKD), Hepatocellular carcinoma (HCC), Obstructive sleep apnoea (OSA), Polycystic ovary syndrome (PCOS) and Chronic Plaque Psoriasis NAFLD is considered the liver manifestation of metabolic syndrome and beyond effects on the liver (risk of cirrhosis and HCC), can also increase the risk of morbidity due to CVD, CKD, psoriasis, PCOS, OSA, and mortality related to T2DM, coronary heart disease, even in absence of well-known risk factors (i.e. smoking, hypertension, T2DM, dyslipidaemia). In this regard, interventions such as lifestyle modification (proper nutrition and exercise), along with pharmacological agents are vital to reduce co-morbidities. Interestingly, the role of the liver seems to be central in the onset and progression of its co-morbidities. However, there are still insufficient information regarding the disease pathways and mechanisms common to these disorders co-occurring with NAFLD.

Within this scenario the appropriate management of NAFLD may have a beneficial effect also on the co-morbidities. At today, the investigation of the common pathogenic mechanisms of the abovementioned inter-related diseases has been approached rather ineffectively, leaving major holes and undermining the development of appropriate management programs for NAFLD/NASH and its related co-morbidities. In order to fill the gap and increase the quality of data for a multi-omic approach we decided to set up a certified local repository. Therefore, the understanding of the pathogenesis of NAFLD and its relevance in the development of related co-morbidities is crucial to guide the development of future treatments and to inform European Union health and economic policies. The clinical impact of NAFLD is considerable and represents a real driver of the major clinical outcomes that impact on the health of the individual, consequently creating a real burden of disease, especially in those populations considered at higher risk of fibrosis such as diabetics or obese. The global burden of NAFLD/NASH and CC require a multi-omic approach in order to prevent and to provide health plans for avoid implications for the population.

Despite the high epidemiology impact, there are still significant areas of unmet clinical need in NAFLD: i) the lack of knowledge on molecular mechanism leading to progression of liver disease; ii) a poor understanding of disease sub-phenotypes; iii) the lack of biomarkers of disease progression that allow risk stratification.

The current availability of the -omics technologies generating libraries of genome-wide data, metabolomes, proteomes and microbiome will allow a precision medicine approach in order to improve the knowledge of disease and to generate a personalized approach to improve the clinical practice and optimize the public health plans for prevention programs and NAFLD management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical phenotype of NAFLD (simple steatosis, NASH, metabolic cirrhosis, NAFLD-HCC) based on any of:
* Liver biopsy providing histological evidence of NAFLD or,
* Biochemical and/or radiological findings consistent with NAFLD
* Average alcohol consumption ≤21/14 units/week (males/females) in preceding 6 months and no history of sustained excessive consumption of alcohol in past 5 years.
* Clearance of HCV infection with new DAAs drugs with a SVR (sustained virological response) period > 6 months
* Presence of risk factors for NAFLD (i.e. diabetes, metabolic syndrome, obesity, psoriasis) and absence of fatty liver at US

Exclusion Criteria:

* Refusal or inability (lack of capacity) to give informed consent.
* Average alcohol ingestion >21/14 units/week (males/females) in preceding 6 months or history of sustained excessive consumption of alcohol in past 5 years.
* History or presence of Type 1 diabetes mellitus.
* Patients not meeting inclusion criteria or judged by the investigator to be unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under the care at Fondazione Policlinico Gemelli IRCCS Hospital
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Registry creation | 35 years
  Set up an observational cohort with NAFLD at different stage of disease (from simple steatosis to cirrhosis and/or HCC)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Rome, Fondazione Policlinico Gemelli IRCCS, Roma, Rome/lazio/italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided